CLINICAL TRIAL: NCT04975802
Title: Effect of Coffeeberry on Mood and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2005
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Mental Fatigue; Alertness; Mood; Cognition
Keywords: alertness; mental fatigue; coffeeberry; coffee fruit
MeSH Terms: conditions — Mental Fatigue | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 mg coffeeberry beverage (Placebo Comparator): Appearance-matched to the other products
  Interventions: Other: Placebo
- 100 mg coffeeberry beverage (Experimental): Appearance-matched to the other products
  Interventions: Dietary Supplement: Coffeeberry
- 300 mg coffeeberry beverage (Experimental): Appearance-matched to the other products
  Interventions: Dietary Supplement: Coffeeberry
- 75 mg caffeine beverage (Active Comparator): Appearance-matched to the other products
  Interventions: Dietary Supplement: Caffeine

INTERVENTIONS:
Other: Placebo — 10 oz (296 ml) cherry flavored still beverage
  Arms: 0 mg coffeeberry beverage
Dietary Supplement: Coffeeberry — 10 oz (296 ml) cherry flavored still beverage
  Arms: 100 mg coffeeberry beverage; 300 mg coffeeberry beverage
Dietary Supplement: Caffeine — 10 oz (296 ml) cherry flavored still beverage
  Arms: 75 mg caffeine beverage

SUMMARY:
The primary aim of this randomised, double-blind, placebo-controlled, cross-over study is to assess the short-term cognitive effects of two beverages containing 100 and 300 mg coffeeberry extract (obtained from the fruit of the coffee plant (Coffea arabica) compared to a placebo beverage. The trial will utilise the COMPASS cognitive assessment system and cognitive demand battery (CDB) and mood visual analogue scales (VAS) with assessments taking place at baseline, 60- and 120-minutes post treatment, on four separate testing days separated by 7 days. A treatment containing 75 mg caffeine will be used as a positive control to document participants' responsiveness to an established psychostimulant.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged 18-49 years, inclusive
* Participants self-report that they are in good health
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial
* Willing to abstain from consumption of caffeine within 12 h of testing
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits
* Willing to refrain from 'over the counter' medications (e.g. pain medication) and stimulant medication for 12 hours, seasonal allergy/hay fever nasal antihistamine medications for 24 hours and oral antihistamines for 48 hours prior to all test visits
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study Investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Current use of prescription medication, except for contraceptives
* Report hypersensitivity to caffeine
* Major trauma or major surgical event within 6 months of screening
* Extreme dietary habits, as judged by the Investigator (high fat, very high protein diets, intermittent fasting, etc.)
* Exposure to coffeeberry within 30 d prior to screening
* History of cancer in the prior two years, except for non-melanoma skin cancer
* Have a visual impairment that cannot be corrected with glasses or contact lenses
* Food allergies/intolerances/sensitivities to any ingredients in the study products (including coffee or related foods/beverages/products)
* Self-report excessive leisure time physical activity (> 7 strenuous bouts per week)
* Have a current or chronic gastrointestinal, sleep, or psychiatric disorders
* Work night shifts or follow a variable work pattern that results in irregular sleep pattern
* Are pregnant, trying to get pregnant or lactating
* Smoke tobacco, vape nicotine or use nicotine replacement products
* Use illegal/recreational drugs
* Unable to demonstrate adequate minimal performance on lab, computer-based cognitive tasks
* Have participated in another clinical trial within past 30 days and/or participation in another PepsiCo trial in the past 6 months
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
* Have learning and/or behavioural disorders such as dyslexia or ADHD
* Excessive caffeine intake (>500 mg per day)
* Have taken dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised)
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Any known active infections
* Does not have a bank account (required for payment)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Mental fatigue Visual Analog Scale (VAS) score | Change from baseline to 120 min post-coffeeberry beverage (100 and 300 mg) consumption during a Cognitive Demand Battery (CDB), compared to placebo beverages. Less mental fatigue is better.
  0-100 mm subjective rating scale, not at all to extremely, within Computerised Mental Performance Assessment framework tasks (COMPASS)
Mental alertness Visual Analog Scale (VAS) score | Change from baseline to 120 min post-coffeeberry beverage (100 and 300 mg) consumption during a Cognitive Demand Battery (CDB), compared to placebo beverages. More mental alertness is better.
  0-100 mm subjective rating scale, not at all to extremely, within Computerised Mental Performance Assessment framework tasks (COMPASS)

SECONDARY OUTCOMES:
Mental fatigue Visual Analog Scale (VAS) score | Change from baseline to 60 min post-coffeeberry beverage (100 and 300 mg) consumption, during a Cognitive Demand Battery (CDB), compared to placebo and caffeine beverages
  0-100 mm subjective rating scale, not at all to extremely, within Computerised Mental Performance Assessment framework tasks (COMPASS). Less mental fatigue is better.
Mental Alertness Visual Analog Scale (VAS) score | Change from baseline to 60 min post-coffeeberry beverage (100 and 300 mg) consumption, during a Cognitive Demand Battery (CDB), compared to placebo and caffeine beverages. More mental alertness is better.
  0-100 mm subjective rating scale, not at all to extremely, from within Computerised Mental Performance Assessment framework tasks (COMPASS)
Motivation Visual Analog Scale (VAS) score | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, during a Cognitive Demand Battery (CDB), compared to placebo and caffeine beverages. More motivation is better.
  0-100 mm subjective rating scale from none to strongest feelings, within Computerised Mental Performance Assessment framework tasks (COMPASS)
Fatigue (Mental State Energy and Fatigue Scales, (EFS)) score | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, following CBD, compared to placebo and caffeine beverages. Less fatigue is better.
  Subjective feelings of mental energy and mental fatigue. Intensity rating scale from none to strongest, yields composite score ranging from 0-300, included within Computerised Mental Performance Assessment framework tasks (COMPASS)
Fatigue (Physical State Energy and Fatigue Scales, (EFS)) score | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, following CBD, compared to placebo and caffeine beverages. Less fatigue is better.
  Subjective feelings of physical energy and physical fatigue. Intensity rating scale from none to strongest, yields composite score ranging from 0-300, included within Computerised Mental Performance Assessment framework tasks (COMPASS)
Alertness (Bond Lader Visual Analog Scale (VAS)) score | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, following CBD, compared to placebo and caffeine beverages. More alertness is better.
  0-100 mm subjective rating scale of intensity of feelings within Computerised Mental Performance Assessment framework tasks (COMPASS)
Calmness (Bond Lader Visual Analog Scale (VAS)) score | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, following CBD, compared to placebo and caffeine beverages. More calmness is better.
  0-100 mm subjective rating scale of intensity of feelings within Computerised Mental Performance Assessment framework tasks (COMPASS)
Contentedness (Bond Lader Visual Analog Scale (VAS)) score | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, following CBD, compared to placebo and caffeine beverages. More contentedness is better.
  0-100 mm subjective rating scale of intensity of feelings within Computerised Mental Performance Assessment framework tasks (COMPASS)
Change in cognitive function measures (Serial subtraction tasks, rapid visual information processing) scores | Change from baseline to 60 and 120 min post-coffeeberry beverage (100 and 300 mg) consumption, compared to placebo and caffeine beverages. Higher scores are better.
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)
Episodic memory tasks (delayed word recall, delayed word recognition, delayed picture recognition) score | Comparison of recollection between coffeeberry beverage (100 and 300 mg), placebo and caffeine beverages to stimuli presented at baseline versus 120 min post-consumption. More recall is better.
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Jackson, PhD, Principal Investigator — Northumbria University Newcastle, UK
Locations (1):
- Brain, Performance and Nutrition Research Centre Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No